CLINICAL TRIAL: NCT00809900
Title: Bioavailability and Metabolism of Anthocyanins Following Acute Cranberry (Vaccinium Macrocarpon)Consumption
Brief Title: Bioavailability and Metabolism of Anthocyanins Following Acute Cranberry Consumption
Status: Completed | Type: Observational
Sponsor: Tufts University (Other)
Responsible Party: Paul E. Milbury, Ph.D., Tufts University
Other Study IDs: Tufts 7903
Record Dates: First submitted 2008-12-15; First posted 2008-12-17 (Estimated); Last update posted 2009-12-02 (Estimated); Status verified 2008-12

CONDITIONS: Bioavailability; Cardiovascular Disease
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Dietary Supplement: Cranberry Juice Consumption
  Interventions: Dietary Supplement: Experimental

INTERVENTIONS:
Dietary Supplement: Experimental — Administration of of 480 mL cranberry juice
  Other Names: Cranberry Juice

SUMMARY:
This study hypothesis is that anthocyanins from cranberry juice are bioavailable and can be measured in blood and urine after a single acute consumption of cranberry juice.

DETAILED DESCRIPTION:
Little is known about the acute or chronic pharmacokinetics and metabolism of anthocyanins consumed in amounts relevant to usual dietary intakes. Thus, we hypothesize that anthocyanins from a single oral dose of cranberry juice will be absorbed quickly and can be measured in the circulation and urine within 2-4 h. Further, these anthocyanins will undergo a degree of metabolism but will circulate as well as be removed from blood as both parent compounds and metabolic products.

This research proposal is submitted as an independent sub-study of an existing project, "Effects of Cranberry Juice on Endothelial Function in Patients with Coronary Artery Disease", conducted by Joseph A. Vita, MD at the Boston University School of Medicine and sponsored by Ocean Spray Cranberries, Inc.

This study includes 15 subjects aged 21-80 y and with demonstrated endothelial dysfunction and angiographically proven coronary artery disease who will receive a single dose of 480 mL cranberry juice.

To test the hypotheses of the study to be conducted at HNRCA Tufts, we will utilize blood and urine samples that are already collected and stored. We will separate and analyze anthocyanins in these samples by HPLC and determine the pharmacokinetics of relevant anthocyanins.

ELIGIBILITY:
Inclusion Criteria:

* Stable CAD Patients
* Men & postmenopausal women
* Aged 21-80 years
* All Ethnic Groups
* English Language

Exclusion Criteria:

* Subjects with heart failure are not eligible for participation in this study.
* Women with a positive urine beta HCG pregnancy test and lactating women or women who are planning to become pregnant.
* Clinical history of other major illness including end-stage cancer, renal failure, hepatic failure, gastrointestinal disorders that may impair absorption, or other conditions that in the opinion of the principal investigator make a clinical study inappropriate.
* Regular use of oral steroids
* Cigarette smoking and/or nicotine replacement use
* Regular daily intake of ≥ 2 alcoholic drinks
* Illicit drug use
* History of a psychological illness or condition such as to interfere with the subject's ability to understand the requirements of the study.
* No dietary supplements containing phenolic compounds, i.e., herbal preparations, or berry containing preparations (such as cranberry capsules) for one month prior to study admission.
* Treatment with an investigational new drug within the last 30 days.

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects aged 21-80 y and with demonstrated endothelial dysfunction and angiographically proven coronary artery disease
Sampling Method: Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2007-06; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
Anthocyanin levels in plasma and urine | 0, 2, and 4 hours

CONTACTS AND LOCATIONS:
Overall Officials: Paul E. Milbury, Ph.D., Principal Investigator — Tufts University
Locations (1):
- Jean Mayer USDA Human Nutrition Center on Aging at Tufts University, Boston, Massachusetts, United States